CLINICAL TRIAL: NCT03562741
Title: Outcomes and Data Collection for Fecal Microbiota Transplantation for the Treatment of Recurrent Clostridium Difficile
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krunal Patel (Other)
Responsible Party: Sponsor-Investigator, Krunal Patel, Principal Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00003682
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-05

CONDITIONS: Clostridium Difficile Infection Recurrence; Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): Subjects receive intervention of stool transplanted to the colon via colonoscopy.
  Interventions: Procedure: Fecal Microbiota Transplantation

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Transplantation of Screened donor stool as part of Fecal Microbiota Transplantation

SUMMARY:
The purpose of this study is to see if stool transplant performed by colonoscopy is effective at treating recurrent Clostridium difficile (C. diff) infection of the colon. During the procedure a stool sample is taken from a healthy donor (usually family member or close friend) and transplanted directly into the colon of the patient with C. diff infection. The goal of this experimental procedure (called fecal microbiota transplantation) is to replenish the good bacteria in the colon that can help prevent C. diff infection from coming back after treatment.

DETAILED DESCRIPTION:
Fecal microbiota transplantation (FMT) involves administering fecal material from a healthy individual into the gastrointestinal tract of the patient. This has been done in the past for recurrent colitis secondary to Clostridium difficile infection (CDI) using different methods such as through nasogastric tube, fecal retention enemas, and by colonoscopy. This method of treatment was introduced over 50 years ago with high success rates, although it has not been until recent that more case studies have been performed, with continued success rates of approximately 90%. Studies have found this therapy to be effective with resolution of symptoms in most patients, and have found it to be both cost effective and safe.

The purpose of this study is to use a standardized published protocol for fecal microbiota transplantation performed by colonoscopy and record the success rate and outcomes of FMT therapy for patients with recurrent CDI at the UMassMemorial Medical Center. In addition, the cost of this therapy will be compared to conventional antibiotic treatment. The reduction in hospitalizations will also be monitored compared with historical controls.

The hypothesis of this study is that FMT therapy will show resolution of infection in most patients with recurrent CDI, with an overall reduction in cost to the hospital for recurrent admissions for Clostridium difficile colitis as compared to historical controls. Historical controls will be defined as patients with recurrent positive Clostridium difficile stool samples treated in the traditional fashion with antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Two or more recurrences of C. difficile infection (CDI) with recurrence defined as a positive test result, e.g. Polymerase Chain Reaction (PCR) test and with appropriate symptoms within 2-8 weeks of last positive result, provided that symptoms from earlier episode resolved with or without therapy.
* Failed standard therapy with oral metronidazole and/or oral vancomycin
* One or more episodes of severe CDI resulting in hospitalization and not responding to standard antibiotic therapy. Hospitalization for CDI occurs in the setting of severe diarrhea, abdominal pain and signs of systemic toxicity

Exclusion criteria:

* Age <16 years old
* patients with acute severe colonic dilation at risk for colonic perforation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-01-16 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2027-01-16 (Estimated)

PRIMARY OUTCOMES:
Clostridium Difficile (C. diff) resolution' | 12 months
  Longterm resolution of C. diff associated diarrhea after Fecal Microbiota Transplantation (FMT) therapy

CONTACTS AND LOCATIONS:
Overall Officials: Krunal Patel, Principal Investigator — UMass Medical School
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No